CLINICAL TRIAL: NCT04825652
Title: Managed Access Program (MAP) Cohort Treatment Plan [CAAA617A12001M] to Provide Access to 177Lu-PSMA-617 for Patients With Metastatic Castration-resistant Prostate Cancer.
Brief Title: 177Lu-PSMA-617 Managed Access Program for mCRPC Patients
Status: No longer available | Type: Expanded Access
Sponsor: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Other Study IDs: CAAA617A12001M
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC)
Keywords: metastatic castration-resistant prostate cancer; mCRPC; 177Lu-PSMA-617
MeSH Terms: interventions — Pluvicto; PSMA-11

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Participants will receive 7.4 GBq (200 mCi) +/- 10% 177Lu-PSMA-617 once every 6 weeks for 6 cycles.
Drug: PSMA-11 — Patients will receive a dose of gallium (68Ga) gozetotide that is 1.8-2.2 MBq/kg of body weight (0.049-0.059 mCi/kg), with a minimum dose of 111 MBq (3mCi) up to a maximum dose of 259 MBq (7 mCi).

SUMMARY:
The purpose of this Cohort Treatment Plan is to allow access to 177Lu-PSMA-617 for eligible patients diagnosed with metastatic castration-resistant prostate cancer (mCRPC). The patient's treating physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

DETAILED DESCRIPTION:
PSMA-11 will be provided in certain cases where it may be required as a diagnostic imaging agent. PSMA-11 is used to confirm the presence of PSMA positive lesions in patients, which then makes them eligible for treatment with 177Lu-PSMA-617.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥ 18 years of age.
2. Patients must have progressive mCRPC. Documented progressive mCRPC will be based on at least 1 of the following criteria:

   * Rising PSA according to PCWG3 criteria (2 rising values above a baseline at a minimum of 1-week intervals) and PSA ≥2.0 ng/mL
   * Soft-tissue progression defined as per prostate cancer working group 3 (PCWG3)-modified RECIST v1.1
   * Progression of bone disease as per PCWG3 criteria
3. Patients must have mCRPC with histological, pathological, and/or cytological confirmation of adenocarcinoma of the prostate.
4. Patients must have ≥ 1 metastatic lesion that is present on baseline CT, MRI, or bone scan imaging.
5. Patients must have prostate-specific membrane antigen (PSMA)- positive prostate cancer, as determined by PSMA-targeted PET / CT scan.
6. Patients must have a castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L).
7. Patients must have received at least one NAAD (such as enzalutamide and/or abiraterone).
8. Patients must have been previously treated with at least 1, but no more than 2 previous taxane regimens. A taxane regimen is defined as a minimum exposure of 2 cycles of a taxane. If a patient has received only 1 taxane regimen, the patient is eligible if:

   a. The patient's physician deems him unsuitable to receive a second taxane regimen (e.g. frailty assessed by geriatric or health status evaluation, intolerance, etc.).
9. Patients must have recovered to ≤ Grade 2 from all clinically significant toxicities related to prior therapies (i.e. prior chemotherapy, radiation, immunotherapy, etc.).
10. Patients must have adequate organ function:

    1. Bone marrow reserve:

       * White blood cell (WBC) count ≥ 2.5 x 10^9/L (2.5 × 10^9/L is equivalent to 2.5 × 10^3/μL and 2.5 × K/μL and 2.5 × 10^3/cumm and 2500/μL) OR absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (1.5 × 10^9/L is equivalent to 1.5 × 10^3/μL and 1.5 × K/μL and 1.5 × 10^3/cumm and 1500/μL).
       * Platelets ≥ 100 × 10^9/L (100 × 10^9/L is equivalent to 100 × 10^3/μL and 100 × K/μL and 100 × 10^3/cumm and 100 000/μL).
       * Hemoglobin ≥ 9 g/dL (9 g/dL is equivalent to 90 g/L and 5.59 mmol/L).
    2. Hepatic:

       * Total bilirubin ≤ 1.5 × the institutional upper limit of normal (ULN). For patients with known Gilbert's Syndrome ≤ 3 × ULN is permitted.
       * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3.0 × ULN OR ≤ 5.0 × ULN for patients with liver metastases.
    3. Renal:

       * Serum/plasma creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min.
       * Albumin > 3.0 g/dL (3.0 g/dL is equivalent to 30 g/L).

Exclusion Criteria:

1. History of hypersensitivity to any drugs or metabolites of similar chemical classes as Lu-PSMA-617.
2. Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy.
3. Transfusion for the sole purpose of making a subject eligible for study inclusion.
4. Patients with a history of central nervous system (CNS) metastases must have received therapy (surgery, radiotherapy, gamma knife) and be neurologically stable, asymptomatic, and not receiving corticosteroids for the purposes of maintaining neurologic integrity.
5. Patients with epidural disease, canal disease and prior cord involvement are eligible if those areas have been treated, are stable, and not neurologically impaired. For patients with parenchymal CNS metastasis (or a history of CNS metastasis), baseline and subsequent radiological imaging must include evaluation of the brain (MRI preferred or CT with contrast).
6. Any pre-existing symptoms, or concurrent severe and/or uncontrolled medical conditions which could compromise safe participation in the MAP.
7. Not able to understand and comply with treatment instructions and requirements.

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Gender Based: Yes — patients diagnosed with metastatic castration-resistant prostate cancer (mCRPC)